CLINICAL TRIAL: NCT05355961
Title: Effect of NorEpinephrine Administration on Ventricular Systolic Function in Septic Shock Patients: the ENESySS Study
Brief Title: Effect of Norepinephrine Administration on Ventricular Systolic Function in Septic Shock
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4774
Record Dates: First submitted 2022-03-23; First posted 2022-05-02 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2022-04

CONDITIONS: Septic Shock
Keywords: NorEpinephrine; Septic Shock; Beta-1adrenergic effect; Ventricular Systolic Function
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples for blood gas analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational, pharmacological, prospective study aims to assess the improvement of ventricular systolic function mediated by norepinephrine (NE) administration in preload non-responders septic shock patients. Left ventricular outflow tract velocity time integral (LVOT-VTI) is an echocardiographic index of ventricular systolic function and it will be measured at different NE dosages.

DETAILED DESCRIPTION:
Norepinephrine (NE) is recommended as first line vasopressor in septic shock. Besides increasing arterial tone and thus arterial pressure, NE improves cardiac output (CO) as a result of two main mechanisms: (i) the increase in venous return due to venoconstriction, in case of preload responsiveness, (ii) the improvement of coronary perfusion through augmentation of diastolic arterial pressure. Experimental data show that NE may incrase cardiac output by exerting also a direct β1-adrenergic stimulation on ventricular myocardial fibers. However, there are few clinical data dealing with the direct effect of NE administration on ventricular systolic function in human septic shock.

Our study aims to demonstrate that norepinephrine administration in early septic shock preload non-responder patients may improve left ventricular outflow tract velocity time integral (LVOT-VTI), measured by trans-thoracic echocardiography (TTE). We will include patients requiring an increase of NE dose for clinical need according to treating physician's decision. For each enrolled patient we will record standard hemodynamic data and perform TTE before NE dosage change (T0). After the increase of NE infusion rate targeting clinical need, a second set (T1) of hemodynamic and TTE data will be obtained.

All TTE examinations will be performed by two experienced and certified clinicians according to current guidelines. After being acquired, all TTE data will be independently analyzed by both clinicians and averaged. LVOT-VTI will be measured in the left ventricular outflow tract on the apical five-chamber (A5C) view. Referring to available literature data, we expect a mean LVOT-VTI of about 18 cm in our patients and we will consider clinically relevant an increase of 15% in LVOT-VTI from T 0 to T 1. We calculated that at least 30 patients need to be enrolled considering an alpha of 0.05 and a power of 80%. The benefits deriving from this study lay in the possibility of improving the clinical understanding of septic shock derived hemodynamic derangements and of widening therapeutic perspectives. Such an information meets the increasing topical need to customize medical interventions, especially in the context of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* less than 6 hours from the diagnosis of septic shock
* ongoing vasopressor therapy by continuous intravenous infusion of norepinephrine
* treating physician's decision to increase norepinephrine dose

Exclusion Criteria:

* preload responsiveness assessed through dynamic indices
* pregnancy
* myocardial disfunction due to active cardiac disease
* inadequate acoustic window for transthoracic echocardiography
* need for emergency treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Preload non-responder patients admitted to the ICU with a diagnosis of septic shock.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Variation of LVOT-VTI | 1 hour
  LVOT-VTI will be measured before and after increasing NE dose. An increase by 15% in LVOT-VTI will be considered clinically relevant.

SECONDARY OUTCOMES:
Variation of left ventricle end-systolic elastance | 1 hour
  Observe the effect of increasing NE infusion rate on left ventricle end-systolic elastance.
Variation of tricuspid annulus plane systolic excursion | 1 hour
  Observe the effect of increasing NE infusion rate on tricuspid annulus plane systolic excursion.
Variation of LVOT-VTI, left ventricle end-systolic elastance and tricuspid annulus plane systolic excursion in patients with pre-existing depressed left ventricular systolic function. | 1 hour
  Observe the effect of increasing NE infusion rate on ventricular systolic function in patients with preexisting depressed left ventricular systolic function defined by a LVEF ≤ 45%.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Carelli, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM, Italy